CLINICAL TRIAL: NCT03572907
Title: Use of Titanium Plate in Rhinoplasty in Patients With Cleft Lip and Palate: Aesthetic and Functional Impact. TROPIC (Titanium RhinOPlasty ImpaCt)
Brief Title: Use of Titanium Plate in Rhinoplasty in Patients With Cleft Lip and Palate : Aesthetic and Functional Impact.
Acronym: PETROL/TROPHIC
Status: Withdrawn | Type: Observational
Why Stopped: Investigators decision
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0328
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-06

CONDITIONS: Cleft Lip; Cleft Palate
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rhinoplasty questionnaire — Each patient will complete a validated rhinoplasty questionnaire (Rhinoplasty Outcome Evaluation) before and after the intervention

SUMMARY:
The patients in this study are all born with a cleft lip and palate. They underwent several interventions in childhood to take care of it.

Professor Gleizal offered them a secondary rhinoplasty aimed at normalizing the appearance of their nose.

In this malformative and multioperated context, typical nasal deformities affect the tip of the nose, which appears to be sagging and asymmetrical. Scarred soft tissues exert an important retractile force against which conventional rhinoplasty techniques often remain insufficient.

The use of columellar struts makes it possible to give again projection to the tip of the nose but when this strut is made from cartilage or bone, it is absorbed with the time. Moreover, these interventions require a remote removal of the site of interest (costal cartilage, tibial crest, calvaria) which generates additional morbidity.

The investigators propose an alternative using a synthetic graft of titanium. This material has been used for many years for its excellent biocompatibility and trauma resistance.

28 patients were able to benefit from this technique between March 1, 2016 and March 1, 2018.

The investigators wish to evaluate the aesthetic and functional results from the patient's point of view by submitting them to one validated rhinoplasty questionnaire after the end of the patient's inclusion.

ELIGIBILITY:
Inclusion Criteria:

* patient over 12 years
* patients with cleft lip and palate operated by Pr Gleizal of a secondary rhinoplasty using a titanium columellar strut
* between January 1, 2016 and March 1, 2018
* patient not having opposed their participation

Exclusion Criteria:

* patient not mastering the French language
* patient participating in interventional research

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cleft lip and palate who underwent secondary rhinoplasty using a titanium columelar strut between March 1, 2016 and March 1, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Rhinoplasty Outcome Evaluation scores | 1 month
  Comparison of pre- and postoperative ROE (Rhinoplasty Outcome Evaluation) scores in patients with cleft lip and palate who benefited from the placement of a titanium columellar strut.
  Each patient completes the questionnaire before and after the intervention. Then the investigators compare these scores to evaluate the improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de chirurgie maxillo-faciale - Hôpital de la Croix Rousse - Groupement Hospitalier Nord - Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No